CLINICAL TRIAL: NCT04704856
Title: Supervised Exercise to Promote Infiltration of NK-cells Into the Tumor
Acronym: SPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Hans J. van der Vliet, MD, PhD, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020.253 NL72539.029.20
Record Dates: First submitted 2020-12-18; First posted 2021-01-12 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Stage I-III breastcancer; Neoadjuvant chemotherapy; Exercise; NK-cells
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventiongroup (Active Comparator): Interventiongroup, undergo supervised exercise for the first 6 weeks.
  Interventions: Behavioral: Supervised exercise
- Controlgroup (No Intervention): Controlgroup, do not undergo supervised exercise for the first 6 weeks (possibility to undergo supervised exercise after 6 weeks).

INTERVENTIONS:
Behavioral: Supervised exercise — Supervised exercise during first 6 weeks of neoadjuvant chemotherapy.
  Arms: Interventiongroup

SUMMARY:
'Supervised exercise to PRomote Infiltration of NK-cells into the Tumor? The objective of this feasibility study is to 1) study trial feasibility in terms of patient enrollment and the percentage of tumor biopsies that can be examined successfully, and 2) generate preliminary data on the potential effects of exercise on immune function assessed in the tumor and in blood.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled feasibility trial, in which 20 women with breast cancer scheduled for neoadjuvant 2 or 3 weekly AC-T(H) chemotherapy will be randomized into a combined aerobic and resistance exercise intervention group or a usual care (no exercise) control group, during the first 6 weeks (2 or 3 cycles) of chemotherapy. Patients from the control group will receive care as usual and are requested to maintain their usual daily physical activities. In order to limit contamination (increase of exercise in the control group), non-participation and prevent dropout, the control group will be offered the same 6-week exercise intervention after the tumor biopsy has been taken after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* stage I-III breast cancer
* scheduled for neoadjuvant chemotherapy with 2 or 3-weekly Adriamycin/Cyclofosfamide, followed by Paclitaxel weekly +/- trastuzumab
* willing to undergo an additional ultrasound guided biopsy
* ECOG-performance score ≤ 2 (able to perform basic activities of daily living such as walking or biking)

Exclusion Criteria:

* addition of immuno- or targeted therapy at start of neoadjuvant chemotherapy
* currently participating in structured vigorous aerobic exercise and/or resistance exercise

(≥2 days per week).

* cognitive disorder or severe emotional instability
* presence of other disabling co-morbidity that might hamper physical exercise e.g. heart failure (NYHA classes 3 and 4), chronic obstructive pulmonary disease (COPD, gold 3 and 4), orthopaedic conditions and neurological disorders (e.g., hernia, paresis, amputation, active rheumatoid arthritis);
* immunosuppressive medication (e.g. corticosteroids (other than used as part of standard chemotherapy premedication protocol), cyclosporine)
* immunodeficiency (primary or secondary)
* impossibility to perform an ultrasound-guided biopsy of the tumor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Stage I-III breastcancer
Enrollment: 20 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Participatient Rate | 6 weeks
  Percentage of patient actually enrolled in the study of all patients who will be screened
Successful Examined Biopsies Rate | 6 weeks
  Percentage of tumor biopsies that can be examined successfully

SECONDARY OUTCOMES:
Generate preliminary data | 6 weeks
  on the potential effects of exercise on immune function (Tumor tissue will be investigated by immunohistochemistry (IHC) to assess immune cell infiltration into the tumor with a specific focus on NK-cell frequency and phenotype) assessed in the tumor and in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Hans van der Vliet, Prof., Principal Investigator — Amsterdam UMC, location VUmc; Laurien Buffart, PhD, Principal Investigator — Radboud University Medical Center; Marieke ten Tusscher, MSc., Study Chair — Amsterdam UMC, location VUmc; Susanne van der Velde, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - Flevoziekenhuis, Almere Stad, Flevoziekenhuis
  - VU Medical Center, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Yes
POLARIS study (PROSPERO 2013 CRD42013003805)
Supporting Information: Analytic Code
Time Frame: 01-01-2023 t/m 01-01-2025
Access Criteria: anonymous

DOCUMENTS (1):
  • Study Protocol (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04704856/Prot_000.pdf